CLINICAL TRIAL: NCT00650871
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Effects of GW679769 (30mg and 90mg) on Sleep Continuity, PSG Sleep Recordings, Subjective Sleep Assessment, and Daytime Cognitive Function in Subjects With Primary Insomnia
Brief Title: A Study to Evaluate the Effects of GW679769 on Sleep and Cognitive Function in Subjects With Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Diagnostic
Other Study IDs: GW679769/903
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: sleep,; polysomnography.; GW679769,; primary insomnia,; cognitive function,
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — casopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW679769
Drug: Placebo
  Other Names: GW679769

SUMMARY:
A study to investigate the effects of GW679769 on sleep and cognition. Potential subjects participate in a clinical screening visit and a two-night PSG recording session in the sleep laboratory. Eligible subjects then participate in three separate two-night PSG sessions in which they are randomized to receive placebo or one of two doses of GW679769 60 minutes prior to bedtime, one treatment for each session in a balanced order. Each treatment session is separated by a two-week drug-free period and occur on the same day of the week. A safety follow-up visit occurs 2 weeks after the last treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects with primary insomnia with normal EG may be eligible for inclusion.

Exclusion Criteria:

* clinically significant physical or psychiatric illness or abnormal sleep patterns.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2004-07-30 (Actual); Primary Completion 2005-08-30 (Actual); Study Completion 2005-08-30 (Actual)

PRIMARY OUTCOMES:
Mean Wake time after sleep onset (WASO) derived from PSG recording | Night 1 and 2 of each treatment period (Approximately up to 31 Days)
  WASO was measured from persistent sleep onset to lights on. It was calculated as number of wake epochs from persistent sleep onset to lights on divided by 2. WASO measures was analyzed using a mixed effect model with session and treatment as fixed effect and participants as random effect.

SECONDARY OUTCOMES:
Mean total sleep time (TST) as objective PSG measures of sleep continuity | Night 1 and 2 of each treatment period (Approximately up to 31 days)
  TST was defined as duration of Rapid Eye Movement (REM) plus non-REM (NREM)(Stage 1, Stage 2, Stages 3/4) sleep from lights off to lights on. It was calculated as number of REM plus NREM (Stage 1, Stage 2, Stages 3/4) epochs from lights off to lights on divided by 2.
Mean latency to persistent sleep (LPS) as objective PSG measures of sleep continuity | Night 1 and 2 of each treatment period (approximately 31 days)
  LPS was measured from lights off to the first epoch of 20 consecutive non-wake epochs (sleep onset).It was calculated as number of epochs from lights off to the first of 20 consecutive non-wake epochs (sleep onset) divided by 2.
Mean wake during sleep (WDS) as objective PSG measures of sleep continuity | Night 1 and 2 of each treatment period (Approximately up to 31 days)
  WDS was the duration, in min, of wakefulness from persistent sleep onset to final epoch of sleep (stage 1, 2, 3/4, or REM), and corresponds to WDS. WDS was defined as duration of wakefulness from persistent sleep onset to final epoch of sleep (stage 1, 2, 3/4 or REM) (min). An awakening was defined as a PSG recording of at least one wake epoch, bracketed by an epoch of stage 1, 2, or stage 3/4 of NREM sleep or REM sleep. The score was derived by a central PSG reader and was analyzed as the mean of the PSG WDS recordings obtained on two consecutive nights.
Mean wake after sleep (WAS) as objective PSG measures of sleep continuity | Night 1 and 2 of each treatment period (Approximately up to 31 days)
  WAS defined as the duration of wakefulness, in min, from final epoch of sleep to lights on The score was derived by a central PSG reader and was analyzed as the mean of the PSG WAS recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used. The overall WAS for night 1 and 2 was reported.
Mean number of 1 minute awakenings during sleep as objective PSG measures of sleep continuity | Night 1 and 2 of each treatment period (Approximately up to 31 days)
  Number of periods of awakening from persistent sleep onset to lights on were recorded. Number of times after persistent sleep onset that there was a wake entry on the PSG recording of at least 1 minute duration (at least 2 consecutive wake epochs). Pairs of awakenings were separated an epoch of NREM sleep or REM sleep. Two wake entries of at least one minute separated by stage 1 sleep was considered as a single awakening.
Total Time in NREM Stage 1 and stage 2 as objective PSG measures of sleep structure | Night 1 and 2 of each treatment period (Approximately up to 31 days)
  NREM sleep time was defined as the duration (in min) of NREM sleep during time in bed. The scores were derived by a central PSG reader and was analyzed as the mean of the PSG NREM recordings obtained on two consecutive nights.Total Time in NREM Stage 1 and stage 2 as objective PSG measures of sleep structure were recorded on night 1 and 2 and mean over the two nights was reported.
Total Time in Slow Wave Sleep (SWS) as objective PSG measures of sleep structure | Night 1 and 2 of each treatment period (Approximately up to 31 days)
  SWS was defined as the duration, in min, of stage 3 or 4 duration during time in bed. Total time in SWS as objective PSG measures of sleep structure was recorded on night 1 and 2 and mean over the two nights was reported.
Total Time in REM as objective PSG measures of sleep structure | Night 1 and 2 of each treatment period (Approximately up to 31 days)
  REM sleep time was also known as stage REM duration. It was defined as the number of minutes of stage REM during time in bed. Time in REM as objective PSG measures of sleep structure was recorded on night 1 and 2 and mean over the two nights was reported.
Latency to REM as objective PSG measures of sleep structure | Night 1 and 2 of each treatment period (Approximately up to 31 days)
  Latency to REM as objective PSG measures of sleep structure was recorded on night 1 and 2 and mean over the two nights was reported.
Total sleep time (TST) as parameter of subjective post-sleep questionnaire | Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  TST was the duration in min of REM plus NREM (Stage 1, Stage 2, Stages 3/4) sleep from lights off to lights on obtained on two consecutive nights of each PSG session. It was calculated as the number of REM plus NREM (Stage 1, Stage 2, Stages 3/4) epochs from lights off to lights on that is during Time in Bed (TIB). TST as parameter of subjective post-sleep questionnaire was recorded in response to the question, How long (total hours and minutes) do you think you slept last night? The questionnaire was reported by the participants on the next day of the PSG nights 1 and 2 and mean over the two nights was reported.
WASO as parameter of subjective post-sleep questionnaire | Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  WASO was defined as the amount of time awake after persistent sleep onset to lights on. An awakening was defined as a PSG recording of at least one wake epoch, bracketed by an epoch of stage 1, 2, or stage 3/4 of NREM sleep or REM sleep. WASO was calculated as summation of number of WAS and number of WDS. WASO as parameter of subjective post-sleep questionnaire was assessed from response of the question Did you wake up during the night? The questionnaire was reported by the participants on the next day of the PSG nights 1 and 2 and mean over the two nights was reported.
Sleep onset latency (SOL) as parameter of subjective post-sleep questionnaire | Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  SOL is the time required to fall asleep. SOL as parameter of subjective post-sleep questionnaire was recorded in response to the question, How long do you think it took you to fall asleep last night? The questionnaire was reported by the participants on the next day of the PSG nights 1 and 2 and mean over the two nights was reported.
Number of awakenings as parameter of subjective post-sleep questionnaire | Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  Number of awakenings was subjective (participant-rated) measurement of number of awakening after sleep onset. Number of awakenings as parameter of subjective post-sleep questionnaire was recorded in response to the question, How many times do you think you woke up? The questionnaire was reported by the participants on the next day of the PSG nights 1 and 2 and mean over the two nights was reported.
Sleep quality (SQ) as parameter of subjective post-sleep questionnaire | Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  SQ as parameter of subjective post-sleep questionnaire was recorded in response to the question, How would you describe the quality of your sleep last night? The responses from participants were recorded as very poor = 1, poor = 2, average= 3,good= 4, very good= 5 indicating the SQ. The questionnaire was reported by the participants on the next day of the PSG nights 1 and 2 and mean over the two nights was reported.
Digit symbol substitution test (DSST) as a measure of daytime cognitive function | Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  DSST was a widely used measure of performance impairment. It is a typical test of association involved in substituting symbols for digits over a period of time. The number of correct signs substituted was taken as the score. Participants marked a geometric pattern associated with one of the digits displayed on a computer screen. Participants had 90 seconds to match as many geometric patterns as possible. The dependent measure were the number of patterns the participant were able to mark correctly (i.e., number of trials correct). Minimum possible score is 0= impaired cognitive function, there was no upper limit of the score. Higher the score indicated betterment in the daytime cognitive function. Mean DSST was calculated from the observations recorded on days followed by first and second PSG nights and mean over the two nights was reported.
Mean Hopkins Verbal Learning Test-Revised (HVLT-R) score including total recall and delayed recall as a measure of Daytime Cognitive Function | Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  HVLT-R assesses verbal learning and memory. It comprised of four subscales including total recall, delayed recall, retention score, and recognition discrimination index. The total recall score was the number of correctly reported words in each of the 3 learning trials and the score ranged from 0 to 36. The delayed recall score was the number of correctly reported words in the delayed recall test and the score ranged from 0 to 12. The retention score represented the score on the delayed recall test divided by the higher of the recall scores from learning trials 2 and 3, multiplied by 100. It was practically ranged from 0 to 100. Higher score indicated betterment in the daytime cognitive function. The recognition discrimination index (RDI) was calculated by subtracting the total false positives score (semantically-related plus semantically un-related) from the total true-positives score obtained in the delayed recognition test).
HVLT-R (Retention %) as a measure of daytime Cognitive Function | Night 1, Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  The HVLT-R offers a brief assessment of verbal learning and memory (recognition and recall) and its use had been validated with brain-disordered populations. Eight distinct forms of the HVLT-R were available, eliminating practice effects on repeated administrations. Each form consists of a list of 12 nouns (targets) with four words drawn from each of three semantic categories. The semantic categories differ across the eight forms, but the forms were very similar in their psychometric properties. The HVLT-R tasks included three learning trials, a delayed recall trial (20-25 minute delay), and a yes/no delayed recognition trial. This latter trial consists of a randomized list that includes the 12 target words and 12 non-target words, 6 of which are drawn from the same semantic categories as the targets. Mean percent retention of the target words was measured as a daytime cognitive function and mean over the three measures recorded at Night 1, Day 1 and 2 are reported.
HVLT-R (Recognition Discrimination Index [RDI]) as a measure of daytime Cognitive Function | Night 1, Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  The HVLT-R offers a brief assessment of verbal learning and memory (recognition and recall) and its use had been validated with brain-disordered populations. Eight distinct forms of the HVLT-R were available, eliminating practice effects on repeated administrations. Each form consists of a list of 12 nouns (targets) with four words drawn from each of three semantic categories. The semantic categories differ across the eight forms, but the forms were very similar in their psychometric properties. The HVLT-R tasks included three learning trials, a delayed recall trial (20-25 minute delay), and a yes/no delayed recognition trial. This latter trial consists of a randomized list that includes the 12 target words and 12 non-target words, 6 of which are drawn from the same semantic categories as the targets. Recognition Discrimination Index of the target words was measured as a daytime cognitive function and mean over the three measures recorded at Night 1, Day 1 and 2 are reported.
Leeds Sleep Evaluation Questionnaire as scales for sleepiness/alertness | Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  LSEQ had been used to monitor subjectively perceived changes in sleep during psychopharmacological investigation involving a variety of psychoactive agents. The questionnaire contains ten self-rating 100-mm-line analogue questions pertaining to four consecutive aspects of sleep: getting to sleep (GTS), QOS, awakening from sleep (AFS) and behaviour following wakefulness (BFW). Scores on the four LSEQ subscales vary between 100 (the largest possible positive change experienced after drug administration) and 0 (the largest possible negative change experienced after drug administration).
Stanford Sleepiness Scale as scales for sleepiness/alertness | Day 1 and 2 post PSG of each treatment period (Approximately up to 31 days)
  Stanford Sleepiness Scale was assessed using the sleep evaluation questionnaire on Day 1 and 7 prior to dosing and at approximately 1 hour intervals after dosing until discharge from the clinic. It was rated on a seven point scale (1-7), where lower score indicates active and higher score indicates sleep onset soon; 1: feeling active, vital, alert, or wide awake, 2: functioning at high levels, but not at peak; able to concentrate, 3: awake, but relaxed; responsive but not fully alert, 4: somewhat foggy, let down, 5: foggy; losing interest in remaining awake; slowed down, 6: sleepy, woozy, fighting sleep; prefer to lie down, 7: no longer fighting sleep, sleep onset soon; having dream-like thoughts and X: asleep. The mean over Day 1 and Day 2 post PSG nights are reported.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania